CLINICAL TRIAL: NCT02085005
Title: Phase II Study of First-line Capecitabine Plus Oxaliplatin Plus Aflibercept for 6 Cycles Followed by Capecitabine Plus Aflibercept as Maintenance Therapy in Patients With Metastatic Colorectal Cancer: DROP and GO Trial
Brief Title: Capecitabine Plus Aflibercept as Maintenance Therapy Following Capecitabine Plus Oxaliplatin Plus Aflibercept in Patients With Metastatic Colorectal Cancer
Acronym: Drop and Go
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS13787; U1111-1149-0237 (Other: UTN)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Capecitabine; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental): Intravenous (IV) infusion on Day 1 every 3 weeks, followed by CAPOX (capecitabine by oral administration on Day 1 to Day 14 and oxaliplatin intravenous (IV) infusion on Day 1 every 3 weeks) for the induction treatment period (6 cycles) after which the patient may enter the maintenance period during which the treatment is Aflibercept + Capecitabine
  Interventions: Drug: Capecitabine; Drug: Aflibercept AVE0005; Drug: Oxaliplatin SR96669

INTERVENTIONS:
Drug: Capecitabine — Pharmaceutical form:tablet Route of administration: oral
Drug: Aflibercept AVE0005 — Pharmaceutical form:concentrate for infusion Route of administration: intravenous
Drug: Oxaliplatin SR96669 — Pharmaceutical form:solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

Efficacy: To assess the progression-free survival rate at 10 months in patients on maintenance therapy with capecitabine plus aflibercept.

Secondary Objectives:

To evaluate:

* Efficacy: Progression Free Survival (PFS)
* Efficacy: Overall Survival (OS)
* Efficacy: Objective Response Rate (ORR) as per Response Evaluation Criteria In Solid Tumors (RECIST version 1.1) criteria
* Health related Quality of Life (HRQL): EORTC QLQ-C30 scores and EQ5D-3L
* Safety

Exploratory Objective:

To collect blood and tumor samples to perform investigations for potential biomarker testing.

DETAILED DESCRIPTION:
Total study duration for a participant can be up to 28 months.

This trial is being conducted in countries where the INN designation for the study molecule is "aflibercept" and this term is therefore used throughout the synopsis. In the US, the US proper name is "ziv-aflibercept".

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years of both sexes
* Histologically confirmed mCRC
* Unresectable metastatic colorectal cancer. (Patient with resectable metastases (liver or lung) is not eligible.)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* A life expectancy of >3 months
* At least one measurable lesion according to RECIST (version 1.1)
* No prior chemotherapy for advanced disease. Patients with prior (neo)adjuvant chemotherapy completed more than 6 months prior metastatic relapse are eligible (adjuvant does not include the chemotherapy after resection of distant metastases).
* Adequate hematological profile (absolute neutrophil count >1.5 x 109/L, platelet count >100 x 109/L, hemoglobin >9 g/dL)
* Adequate liver function: AST, ALT <3.0 x ULN (or <5 xULN in the case of liver function abnormalities due to underlying liver metastases); Alkaline Phosphatase <3 x ULN (or <5 x ULN if due to underlying liver metastases); Total bilirubin <1.5 x ULN
* Serum creatinine < 1.5 x upper limit of normal (ULN). If creatinine 1.0-1.5 x ULN, creatinine clearance will be calculated according to the CKD-EPI formula and creatinine clearance < 60 mL/min will exclude the patient
* Proteinuria <2+ functions
* Signed patient informed consent before beginning specific protocol procedures
* Ability to comply with protocol requirements

Exclusion criteria:

* Less than 4 weeks from prior radiotherapy to the time of inclusion (less than 2 weeks in case of palliative RT on single bone lesion only)
* Less than 4 weeks following major surgery to the time of inclusion or until the surgical wound is fully healed whichever came later (48 hours in case of minor surgical procedure or until wound full healing observed)
* Treatment with any other investigational product within 28 days prior to inclusion
* Other prior neoplasm. Adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or any other cancer from which the patient has been disease-free for > 5 years are allowed
* History of brain metastases (unless adequately controlled, i.e. previously irradiated, inactive brain metastases not requiring active treatment like steroids or antiepileptics), active seizure disorder, uncontrolled spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease
* Any of the following within 6 months prior to inclusion: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack
* Any of the following within 3 months prior to inclusion: Grade 3-4 gastrointestinal bleeding/hemorrhage (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event
* Occurrence of deep vein thrombosis within 4 weeks, prior to inclusion
* Any severe acute or chronic medical condition, which could impair the ability of the patient to participate in the study or interfere with interpretation of study results. Known Acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease requiring antiretroviral treatment
* Pregnant or breast-feeding woman. Positive pregnancy test (serum or urine β-HCG) for women of reproductive potential
* Patient with reproductive potential (M/F) who do not agree to use accepted and effective method of contraception during the study treatment period and for at least 6 months after the completion of the study treatment. The definition of "effective method of contraception" will be based on the Investigator's judgment
* Patient on anticoagulant therapy with warfarin (coumarin-derivative). Anticoagulation with low molecular weight heparin (LWMH) is permitted
* Symptomatic peripheral sensory neuropathy grade ≥ 2 (NCI-CTCAE v4.03)
* Inability to take oral medications
* Prior history of chronic enteropathy, inflammatory enteropathy, chronic diarrhea, malabsorption syndrome, unresolved bowel obstruction/sub-obstruction, surgery more extensive than hemicolectomy, extensive small intestine resection with chronic diarrhea.
* History of hypersensitivity to fluoropyrimidines or known/suspected allergy to any agent given during the study or to any excipient to study drugs
* Known dihydropyrimidine dehydrogenase deficiency
* Any contraindication to administer oxaliplatin, 5-FU, folinic acid or capecitabine as per package insert of each drug
* Uncontrolled hypertension (defined as BP > 140/90 mmHg or systolic BP >160 mmHg when diastolic BP < 90 mmHg, on at least 2 repeated determinations on separate days, or upon clinical judgment) within 3 months prior to study inclusion
* Evidence of clinically significant bleeding diathesis or underlying coagulopathy (e.g. INR>1.5 without vitamine K antagonist therapy), non-healing wound
* History of hypersensitivity to Aflibercept (in case of prior administration for an indication other than cancer, i.e. ophthalmic indication)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival rate at 10 months (PFS@10m) | every 9 weeks, up to 28 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) - Time | every 9 weeks, up to 28 months
Overall Survival (OS) - Time | every 9 weeks, up to 28 months
Assessment of Objective Response Rate (ORR) | every 9 weeks, up to 28 months
Total Score as a measure of Health Related Quality of Life | every 3 weeks, up to end of treatment
Number of participants with adverse events | up to 30 days after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi